CLINICAL TRIAL: NCT00837044
Title: An Evaluation of Treximet in the Treatment of Acute Migraine Headache: A Placebo-Controlled, Double-Blind, Crossover Study, Assessing Cognitive Function.
Brief Title: Treximet in Acute Migraine Headache: Assessing Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurological Research Center (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Keith R. Edwards, M.D., The Neurological Research Center, Inc
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 112488
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Migraine Headache; Cognitive Impairment
MeSH Terms: conditions — Migraine Disorders; Cognitive Dysfunction | interventions — sumatriptan-naproxen; Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Treximet, cognitive testing
  Interventions: Drug: Treximet
- 2 (Placebo Comparator): Placebo, Cognitive testing
  Interventions: Drug: Migraine rescue medication of choice

INTERVENTIONS:
Drug: Treximet — Treximet
  Other Names: Sumatriptan succinate 85mg/Naproxen Sodium 500mg
  Arms: 1
Drug: Migraine rescue medication of choice — Migraine rescue medication of choice
  Arms: 2

SUMMARY:
Migraine headache occurs frequently in women more than men and is associated with symptoms not only of significant pain but also of symptoms typically including of photophobia, phonophobia, nausea and vomiting. Many migraine patients report difficulty in cognition from lack of concentration, difficulty in word finding or inability to remember. Many of these cognitive symptoms seem to be independent of the pain intensity and may occur completely separately from the headache pain but can be disabling. It is likely that the frequency and importance of cognitive symptoms associated with migraine are underreported.

The Mental Efficacy Workload Test (MEWT) is a computerized battery that is designed to be an efficient and accurate measure of cognition during migraine headache. Treximet is a new migraine treatment recently FDA approved for the treatment for the relief of acute migraine that may be effective for the cognitive symptoms for migraine patients who have a history of cognitive dysfunction during a migraine headache. The primary efficacy parameter is to evaluate the effectiveness of treatment with Treximet versus placebo in patients with acute migraine headache measuring neuropsychological function using the MEWT during the migraine and comparing that score with a prior MEWT score when the patient had no migraine symptoms. A double blind, placebo-controlled, crossover study was chosen so that each patient may be her or his own control.

It is the intent of this study to determine the type and intensity of cognitive dysfunction associated with migraine headache and to what extent that Treximet may relieve the cognitive dysfunction in a safe and effective manner.

DETAILED DESCRIPTION:
Overall Study Design:

This study is to be a double blind crossover comparison study in patients during a migraine headache attack, with assessments at one and two hours after treatment. Patients with an IHS diagnosis of migraine with or without aura may be included. The patients will complete a questionnaire regarding the nature of their migraine attacks, including their impression of cognitive impairment if any. Historically associated symptoms will be listed. Menstrual associated migraine history will be assessed. 30 patients will be randomized to Treximet or placebo in a 1:1 manner for the first treatment and in reverse order for treatment on the second migraine attack. In this manner, each patient will be his or her own control. 60 migraine headaches will be treated in this study. Also, it has been previously discussed that after 3 practice sessions with the MEWT, further administration of the MEWT does not produce bias by a practice effect as the ANAM has been shown not to produce bias by a practice effect.10 Therefore, patients will have 3 practice sessions in the clinic before taking the baseline MEWT.

During the baseline period, while the patient is without any migraine symptoms and feeling well (interictal period), three practice trials on the MEWT will be performed and a fourth MEWT trial will be taken with the score recorded for a neuropsychological baseline. When the patient experiences a migraine headache, the patient will rate headache severity and associated symptoms and then take Treximet or matching placebo. The patient will repeat headache and associated symptom checklist and the MEWT at 1 and 2 hours after treatment. Rescue medication will be allowed at 2 hours for those patients who require it.

4.0 Clinical Methods:

4.1 Selection of Study Population:

4.2 Visit 1 (Screen visit): After informed consent reviewed and signed, inclusion and exclusion criteria reviewed and the patient approved for the study, patients will have assessments and practice MEWT sessions as listed below. The patients will then be scheduled for visit 2 .

These assessments will be completed in the following order:

1. . Type(s) of migraine including menstrual migraine
2. . Medical and surgical history
3. . Migraine history: age of onset, age of onset of cognitive dysfunction
4. . Family history of migraine
5. . Prior treatment for migraine, both rescue and preventative
6. . Age, sex, educational background
7. Concomitant medications
8. General physical and neurological examinations
9. Reviewing with patient headache severity and symptom assessment forms
10. Two practice sessions on the MEWT

    4.3 Visit 2 Patient is to return to clinic within 2 weeks to review headache severity and symptom forms to be filled out at home or work while experiencing a migraine. Two MEWT sessions will be taken, one last session for practice and the other for a baseline test to be compared to MEWT assessment while experiencing a migraine. Subject is randomized to treximet or placebo and given medication package and instructions .* Subject is also given MEWT device to take home along with assessments and diary.

    4.4 Visit 3 (Post-treatment visit #1): The patient is to return to the clinic within one week of treating a migraine to review headache severity and symptom assessment forms, MEWT scoring and adverse event (AE) dairy. Patient given second medication package for second migraine treatment.* Subject given MEWT device and assessment forms to take home and complete when experiencing headache.

    4.5 Visit 4 (Post-treatment visit #2): The patient is to return to the clinic within one week of treating the second migraine to review headache severity and symptom assessment forms, MEWT scoring and AD dairy.

    * Patients may take rescue medication of choice after 2 hours of taking Treximet or placebo if they wish.

    5.0 Adverse Events

    An adverse event definition for this protocol is as follows:

    Any unexpected, untoward medical occurrence that is considered clinically significant by the investigator.

    All adverse events fitting this description will be captured and recorded on the case report forms.

    In the event that a subject is withdrawn from the study because of an adverse event, it must be recorded on the CRF as such. The subject should be followed and treated by the investigator until the abnormal parameter or symptom has resolved or stabilized.

    All adverse events will be recorded in the Case Report Form (CRF)

    6.0 Serious Adverse Events

    A serious AE means any adverse event fitting the description above but also containing one of the following:
    * Death
    * Life threatening experience which places the subject at immediate risk of death from the event as it occurred.
    * Full Inpatient hospitalization or prolongation of hospitalization
    * Persistent or significant disability/incapacity
    * Congenital anomaly or birth defect

    Any reports of these events during the conduct of the study will immediately be reported to the sponsor, to the IRB and to Medwatch.

    7.0 Statistical analysis plan, sample size justification and power analysis

    Cognitive function and efficacy analysis (pain relief) will be calculated on the intent-to-treat (ITT) population. Statistics will be presented for headache response (0-3 scale), pain-free response, safety and demographics. Five subsets of MEWT will be used (CPT, MTS, MP, PRT and SRT -see Table 1). Four of the subset tests of the MEWT (CPT, MTS, MP, and PRT) will be scored for 'throughput,' which is the number of correct responses per minute. This is a measure of efficacy that combines both speed and accuracy in a single score. SRT will be calculated for reaction time in msec. Group means will be calculated from each patient's mean for each MEWT subtest and compared to each stage of the migraine: migraine-free, migraine pre-treatment (time zero) and migraine post-treatment (time 1 and 2 hours). Each MEWT subtest will be calculated using a repeated measure 1 x 3 (each stage of migraine: migraine free, pre and post-treatment) by analysis of variance (ANOVA) for statistical significance of at least p = 0.05 or better.

    8.0 Duration of study

    Nine months (30 patients with baseline practice sessions, treatment of 2 separate migraine headaches)

    9.0 Specific drug supply requirements

    Treximet and matching placebo

    10.0 Publication/presentation plan

    Submission to a national and/or international headache meeting as soon as the data have been analyzed. Submission to a peer review journal within 6 months of study analysis completion.

    11.0 Source Documentation and Case Report Form Completion

    Source documents are defined as original documents, data and records. These may include hospital records, clinical and office charts, lab results, cognitive data and information, etc. The Case Report Form documents will serve as the source records for this trial. All forms will be completed within 5 business days of the study visit. A CRF will be provided for each enrolled study subject. All CRFs will be completed using black ink. All corrections will be made by striking through with a single line and writing correct data above, beside, or below the erroneous data, so as not to obscure the original entry. Each correction will be initialed and dated by the person making the correction.

    12.0 Retention and Availability of Records

    The investigator will maintain adequate records for the protocol including signed Informed consents, patient information sheets, completed source documents, CRF's, Lab reports, Medical records, AE reports and information regarding all subjects who discontinued.

    13.0 Ethics

    Good Clinical Practice (GCP) requires that the clinical protocol, any protocol amendments, the Investigators Brochure if applicable, informed consent/assent, and all other forms of subject information related to the study (including advertisements) be reviewed by the IEC/IRB. IRB approval is mandatory before initiating of any study related activities.

    The study will be conducted per the protocol, in accordance with ICH guidelines, applicable regulations, and guidelines governing clinical study conduct and the ethical principles that have their origin in the Declaration of Helsinki.

    14.0 Use of Information/Confidentiality

    All information obtained during the conduct of this clinical trial is considered confidential. This information may be disclosed as deemed necessary by Neurological Research Center Inc or GlaxoSmithKline, Inc. to other clinical investigators, the IEC/IRB, the FDA and other governmental agencies. Patient identifiers will include patient assigned number, age, and sex. Patient Initials will not be released to the company as this is irrelevant information. The investigator will maintain a confidential subject identification code list of all subjects enrolled in the study by name and subject number. This list will be maintained at the investigative site.

ELIGIBILITY:
Inclusion Criteria:

1. Females and male subjects, ages 18-65 inclusive
2. Have migraines with or without aura as expressed by the International Headache Society (IHS) criteria for at least six months and at least one attack per month for three months prior to screening
3. If female, have an acceptable method of contraception during the study, have no plans to become pregnant and have a negative urine pregnancy test at screening and throughout the study.
4. Must be able to follow study protocol including all neuropsychological testing, MEWT assessments and evaluation forms.
5. Must be willing and able to provide written informed consent

Exclusion Criteria:

1. Have more than 15 headache days per month
2. Have hemiplegic or secondary headaches
3. Have significant risk factors for cardiovascular or cerebrovascular disease as assessed by the investigator
4. Are taking any medication that is contraindicated with a triptan or NSAIDs
5. Have any significant concomitant disease
6. Have any allergy to triptans, aspirin or NSAIDs
7. Have a history of substance abuse, psychiatric illness in the last 5 years
8. Are participating or have participated in an investigational drug trial within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-07 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of treatment with Treximet versus placebo in patients with acute migraine headache on the neuropsychological function before treatment and at one and two hours after treatment of a migraine. | 2 hours post dose

SECONDARY OUTCOMES:
To assess incidence and types of neuropsychological deficits by MEWT in patients with acute migraine headache before treatment. | 2 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Edwards, M.D., Principal Investigator — The Neurological Research Center, Inc.
Locations (1):
- The Neurological Research center, Inc, Bennington, Vermont, United States

REFERENCES:
- [Background] Ardila A, Sanchez E. Neuropsychologic symptoms in the migraine syndrome. Cephalalgia. 1988 Jun;8(2):67-70. doi: 10.1046/j.1468-2982.1988.0802067.x. PMID 3401918
- [Background] Stewart WF, Lipton RB, Celentano DD, Reed ML. Prevalence of migraine headache in the United States. Relation to age, income, race, and other sociodemographic factors. JAMA. 1992 Jan 1;267(1):64-9. PMID 1727198
- [Background] Palmer JE, Chronicle EP. Cognitive processing in migraine: a failure to find facilitation in patients with aura. Cephalalgia. 1998 Apr;18(3):125-32. doi: 10.1046/j.1468-2982.1998.1803125.x. PMID 9595204
- [Background] Farmer K, Cady R, Bleiberg J, Reeves D. A pilot study to measure cognitive efficiency during migraine. Headache. 2000 Sep;40(8):657-61. doi: 10.1046/j.1526-4610.2000.040008657.x. PMID 10971662
- [Background] Farmer K, Cady R, Bleiberg J, Reeves D, Putnam G, O'Quinn S, Batenhorst A. Sumatriptan nasal spray and cognitive function during migraine: results of an open-label study. Headache. 2001 Apr;41(4):377-84. doi: 10.1046/j.1526-4610.2001.111006377.x. PMID 11318884
- [Background] Farmer K, Cady R, Reeves D, Bleiberg J. Cognitive efficiency following migraine therapy. In: J. Olsen, T.J. Steiner, R.B. Lipton (Eds.) Reducing the burden of headache: Frontiers in headache research (pp 46-51) New York: Oxford University Press 2003
- [Background] Cernich A, Reeves D, Sun W, Bleiberg J. Automated Neuropsychological Assessment Metrics sports medicine battery. Arch Clin Neuropsychol. 2007 Feb;22 Suppl 1:S101-14. doi: 10.1016/j.acn.2006.10.008. Epub 2006 Nov 21. PMID 17118625
- [Background] Wilken JA, Sullivan CL, Lewandowski A, Kane RL. The use of ANAM to assess the side-effect profiles and efficacy of medication. Arch Clin Neuropsychol. 2007 Feb;22 Suppl 1:S127-33. doi: 10.1016/j.acn.2006.10.007. Epub 2006 Nov 20. PMID 17116387
- [Background] Wilken JA, Kane R, Sullivan CL, Wallin M, Usiskin JB, Quig ME, Simsarian J, Saunders C, Crayton H, Mandler R, Kerr D, Reeves D, Fuchs K, Manning C, Keller M. The utility of computerized neuropsychological assessment of cognitive dysfunction in patients with relapsing-remitting multiple sclerosis. Mult Scler. 2003 Mar;9(2):119-27. doi: 10.1191/1352458503ms893oa. PMID 12708806
- [Background] Roebuck-Spencer T, Sun W, Cernich AN, Farmer K, Bleiberg J. Assessing change with the Automated Neuropsychological Assessment Metrics (ANAM): issues and challenges. Arch Clin Neuropsychol. 2007 Feb;22 Suppl 1:S79-87. doi: 10.1016/j.acn.2006.10.011. Epub 2006 Nov 21. PMID 17118623
- [Derived] Edwards KR, Rosenthal BL, Farmer KU, Cady RK, Browning R. Evaluation of sumatriptan-naproxen in the treatment of acute migraine: a placebo-controlled, double-blind, cross-over study assessing cognitive function. Headache. 2013 Apr;53(4):656-64. doi: 10.1111/head.12052. Epub 2013 Feb 13. PMID 23406052